CLINICAL TRIAL: NCT06920472
Title: Xerogenic Potential of the Most Frequently Prescribed Psychiatric Drugs
Brief Title: This Present Study Can be Used by Clinicians Who Treat Psychiatric Patients: Dentists Might Expect Xerogenic Side Effects of Specific Psychiatric Drugs Which Can Affect Dental Treatment, and the Results Can Help Psychiatrist to Choose the Less Xerogenic Psychiatric Medication
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Other Study IDs: ETT-TUKEB 55/2013
Record Dates: First submitted 2025-01-15; First posted 2025-04-09 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-01

CONDITIONS: Psychiatric Disorders; Xerostomia Due to Hyposecretion of Salivary Gland
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the effects of psychiatric drug therapies on intra- and extra-oral sicca symptoms and salivation. The main question that it aims to answer is:

Does taking psychiatric medication cause oral dryness and/or any changes on whole and minor saliva secretion? Participants taking psychiatric medication answered a 16-question questionnare, and their saliva production was measured by Periotron device and by spitting method.

ELIGIBILITY:
Inclusion Criteria:

In the psychiatric group, the inclusion criteria was taking specific psychiatric medications.

Exclusion Criteria:

In the control group the exclusion criteria was reporting any diseases and taking medicines.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Outpatient Clinic, Department of Psychiatry and Psychotherapy and Dental Teaching Center, Semmelweis University, Budapest, Hungary
Sampling Method: Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Unstimulated whole saliva flow rate (UWS) | through study completion, an average of 1 year
  UWS was determined using the "spitting" method (Sreebny 2000). Whole saliva was collected for 5 minutes into a previously weighted empty cup, and then measured again after collecting the saliva. The results are in ml/min.
Minor salivary gland (MSG) secretions | Through study completion, an average of 1 year
  Palatal and labial MSG flow rates were measured by the Periotron 8010® (Oraflow Inc. Amytiville, USA) device with filter paper discs. The results are transferred into µl/cm2/min.